CLINICAL TRIAL: NCT06847061
Title: Decreasing Disparity in Lung Disease: Pulmonary Rehabilitation for Rural Patients With COPD
Brief Title: Pulmonary Rehabilitation for Rural Patients With COPD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Roberto P. Benzo, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-008332; 1R01NR021634-01 (NIH)
Record Dates: First submitted 2025-02-21; First posted 2025-02-26 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: This study design is control/Wait.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Group (Experimental): Subjects randomized to the treatment arm will begin the home-based pulmonary rehabilitation intervention immediately.
  Interventions: Behavioral: Pulmonary rehabilitation program
- Waitlist Control (Experimental): Subjects randomized to the waitlist control (usual care) arm will be offered the home-based pulmonary rehabilitation intervention after completing the 12-week control period.
  Interventions: Behavioral: Pulmonary rehabilitation program

INTERVENTIONS:
Behavioral: Pulmonary rehabilitation program — Participants are expected to engage in the home-based pulmonary rehabilitation routine at least 24 minutes a day, five to six days a week for the entire 12-week study period.
  The pulmonary rehabilitation routine begins with slow upper body and timed breathing exercises, followed by two slow balance walks for 6 minutes each. The total exercise time again is 24 minutes, followed by a 4-minute mindful breathing meditation/cool down

SUMMARY:
The purpose of this study is to test the uptake, effectiveness, and patient-caregiver-provider experience of a crucial treatment not provided in rural areas: pulmonary rehabilitation.

ELIGIBILITY:
Inclusion Criteria

* 40 years of age or older
* Physician-diagnosed COPD
* Living in a rural area defined by Rural-Urban Commuting Area Codes 4-10
* mMRC score>=1
* English Speaking

Exclusion Criteria

* Inability to walk (orthopedic/neurologic/cardiac limitation causing immobility)
* Cognitive impairment or inability to understand and follow instructions.
* Patients with no COPD symptom burden, no breathlessness (mMRC score 0), as based on our previous studies they usually perceive no benefit from PR and do not have compliance with PR.
* Traditional center-based PR was completed within 3 months of initial study recruitment.
* Transition to hospice or end-of-life care at the time of screening.
* Acute exacerbation at the time of screening.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2029-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Change Chronic Respiratory Questionnaire Physical and Emotional (CRQ-SAS) summary scores | Baseline, 3 months
  The Chronic Respiratory Disease Questionnaire is a 20 item questionnaire assessing the quality of life for patients with chronic obstructive pulmonary disease (COPD).
  The CRQ covers four domains: dyspnea, fatigue, emotional function, and mastery. Questions are scored on a 7-point Likert scale, with 1 representing 'All of the time' and 7 representing 'None of the time'. Higher scores indicate better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Benzo, M.D., Principal Investigator — Mayo Clinic; Teng Moua, M.D., Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials